CLINICAL TRIAL: NCT03471546
Title: Model of Early Palliative Care Intervention in Patients With Newly Diagnosed WHO Grade IV Malignant Glioma, a Single Arm Feasibility Study
Brief Title: Early Palliative Care Intervention in Malignant Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00091481
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-06

CONDITIONS: Malignant Glioma
Keywords: Palliative Care; Pro00091481; Malignant Glioma; Katherine Peters; David Casarett
MeSH Terms: conditions — Glioma | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Patients newly diagnosed with World Health Organization (WHO) Grade IV malignant glioma will be referred to a Palliative Care provider in the clinic, in order to assess the impact of early palliative care intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palliative care (Experimental): Newly diagnosed patients will be referred to a palliative care provider in the clinic for initial consultation and follow-up during their initial treatment for WHO Grade IV malignant glioma. Patients will be asked to complete a number of questionnaires and assessment forms at different time intervals during the course of their initial treatment. In addition, we will ask patients' neuro-oncology providers for feedback regarding their satisfaction with the Palliative Care services provided to the patient.
  Interventions: Behavioral: Palliative Care

INTERVENTIONS:
Behavioral: Palliative Care — Initial consultation and follow-up with a palliative care provider

SUMMARY:
The purpose of this research study is to determine the feasibility and acceptability of incorporating palliative care into the clinical care plans of patients newly diagnosed with malignant brain tumors. Palliative Care is a field of medicine that focuses on providing relief from symptoms and stress related to serious illnesses. This study will assess the feasibility of conducting a future study, and will gather data upon which to appropriately tailor the intervention and the future study design. The statistical analysis of this study will describe 8 components that encompass each of the 4 areas of focus or "domains": acceptability, demand, implementation, and integration.

DETAILED DESCRIPTION:
Patients who agree to participate at their initial consultation in our clinic will receive a referral to a Palliative Care (PC) provider who is also located in our clinic and an initial appointment will be scheduled with the PC provider. The frequency of follow-up visits with the PC provider will be at the discretion of the PC provider and the patient. Visits with the PC and neuro-oncology providers will be scheduled on the same day whenever possible. As part of the study, participants will be asked to complete a number of questionnaires and assessment forms at different time intervals. These questionnaires and assessments are intended to track symptoms experienced during the course of treatment. Total study duration is about nine months.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patient must have histologically confirmed, newly diagnosed WHO grade IV malignant glioma (confirmation from biopsy, sub-total, or gross-total resection)
* Tumor must be de novo grade IV malignant glioma (i.e. NOT transformed from a lower grade)
* Patient should be planning to receive standard chemoradiation (3 or 6 week protocols are acceptable)
* Treating neuro-oncologist agrees to the patient's participation in this clinical trial
* Patient should be able to read and write English

Exclusion Criteria:

* Patient who currently has a PC provider and/or is receiving hospice care or plans on initiating hospice at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Acceptability: Patient satisfaction | 8 months
  Mean scores obtained from patient-completed FAMCARE-P16 questionnaires. The FAMCARE-P16 measures patient satisfaction using 16 items on a Likert scale which are summed together to produce an aggregate score of satisfaction. It will be administered at study completion or when a patient is discharged to hospice or withdraws study participation.
Acceptability: Provider satisfaction | 8 months
  The percentage of providers who respond "Always" or "Most of the time" to the question "Were you satisfied with your patient's care are the palliative care clinic?" among those providers who complete the Palliative Care Clinic (PCC) Referring Provider Satisfaction Survey upon each patient's study completion.
Acceptability: Continuation of follow-up with palliative care provider after initial consultation | 8 months
  The percentage of patients who continue to follow up with their palliative care provider after initial consultation among those who receive initial consultation.
Acceptability: Continuation of follow-up with palliative care provider beyond study period | 8 months
  The percentage of patients who respond "Yes" to the question "Do you plan to continue to see a palliative care provider after your participation on the study is complete?" among those who complete the end of study questionnaires. This question will be included in the questionnaires administered at study completion.
Demand: Time to enroll 50 patients | 2 years
  The difference in months between the date the first patient is enrolled and the date the 50th patient is enrolled.
Demand: Enrollment percentage | 2 years
  The percentage of patients who choose to enroll in the study among those to which the study is offered.
Implementation: Study completion percentage | 2 years
  The percentage of patients who complete all study-related questionnaires and procedures among those enrolled.
Integration: Provider perception of feasibility | 2 years
  The percentage of providers who respond "Yes" or "Yes with modification" to the question "Do you think that this model of early palliative care referral is feasible to integrate into the existing clinical infrastructure in your outpatient oncology clinic?" among those providers who complete the PCC Referring Provider Satisfaction Survey upon each patient's study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — The Preston Robert Tisch Brain Tumor Center; David Casarett, MD, MA, Principal Investigator — Palliative Care
Locations (1):
- The Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/